CLINICAL TRIAL: NCT04083053
Title: High-Resolution Anoscopy Perceived Discomfort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00059426
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Pain; Anal Cancer
Keywords: anoscopy; screening; perianal examination
MeSH Terms: conditions — Pain; Anus Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perianal Exam First (Experimental): Perianal exam that is a part of anal cancer screening will be performed prior to the intraanal portion of the exam (high-resolution anoscopy with biopsy).
  Interventions: Procedure: Perianal Exam; Procedure: high-resolution anoscopy (HRA) with biopsy
- Perianal Exam Last (Experimental): Perianal exam that is a part of anal cancer screening will be performed after the intraanal portion of the exam (high-resolution anoscopy with biopsy).
  Interventions: Procedure: Perianal Exam; Procedure: high-resolution anoscopy (HRA) with biopsy

INTERVENTIONS:
Procedure: Perianal Exam — Perianal Exam is part of anal cancer screening. The perianal skin is also examined under magnification and, less commonly, perianal biopsies are obtained.
Procedure: high-resolution anoscopy (HRA) with biopsy — The HRA exam involves insertion of a plastic anoscope 4-6 cm into the anal canal, with use of 5% acetic acid and Lugol's iodine to highlight abnormal lesions for biopsy. The entire squamocolumnar junction is visualized during the exam, which lasts between 5 and 20 minutes.

SUMMARY:
Study should determine if performing the less uncomfortable part of the exam (the perianal exam) results in less recalled discomfort if performed last vs. if performed first.

DETAILED DESCRIPTION:
Performance of the perianal examination at the end of the high resolution anoscopy (HRA) procedure will lead to patients reporting less discomfort directly following the procedure. The study team hypothesizes at least a 10% decrease in subsequently rated pain scores in the group where the perianal exam is performed last compared to the group where it is performed first.

ELIGIBILITY:
Inclusion Criteria:

* Present for a previously scheduled high resolution anoscopy procedure
* Able to participate in an English written survey following the HRA procedure

Exclusion Criteria:

* Undergoing ablation during the HRA procedure
* Inability to tolerate or complete the HRA procedure
* Unwillingness or inability to complete the post-procedure survey
* Previous participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
High Resolution Anoscopy (HRA) discomfort scale | following the HRA procedure at day one
  Visual analogue scale ranging from 1 to 10 with higher score denoting more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Barroso, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT04083053/ICF_000.pdf